CLINICAL TRIAL: NCT05853913
Title: Impact of Acute Exercise on Brain Insulin Sensitivity in Middle-aged to Older Adults
Brief Title: Acute Exercise on Brain Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Steven K Malin, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022001842
Record Dates: First submitted 2023-04-19; First posted 2023-05-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Aging; Obesity; Insulin Resistance; Cognition; Cardiovascular Disease Risk
Keywords: Exercise
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals will perform both rest and exercise conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rest (No Intervention): Individuals will rest for about 1 hour in the seated position to mimic time exercising.
- Exercise (Experimental): Individuals will exercise for at medium to hard intensity for 1 hour.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise will be walking/jogging at a medium to hard intensity for 1 hour.
  Arms: Exercise

SUMMARY:
Dementia is a leading cause of death in the United States among aging adults. Brain insulin resistance has emerged as a pathologic factor affecting memory, executive function as well as systemic glucose control. Regular aerobic exercise decreases Alzheimer's Disease (AD) risk, in part, through changes in brain structure and function. However, there is limited data available on how exercise impacts brain insulin resistance in aging. This study will test the effect of acute exercise on brain insulin sensitivity in middle-aged to older adults. The study will also examine cognition and cardiometabolic health in relation to brain insulin sensitivity.

DETAILED DESCRIPTION:
Obesity, hypertension, high blood glucose (e.g. prediabetes/type 2 diabetes), and physical inactivity is thought to worsen brain insulin resistance and reduce cerebral blood flow. This suggests lifestyle approaches may be necessary to counteract declines in brain health. Regular aerobic exercise decreases Alzheimer's Disease (AD) risk, in part, through changes in brain structure and function. Moreover, exercise-related structural changes in the brain, namely increased hippocampal volume, is linked to improved memory. However, there is limited data available on how exercise impacts brain insulin resistance in aging. It is also unclear if one bout of exercise may help improve brain insulin responses to insulin before fitness gains or weight loss in people at risk for dementia, type 2 diabetes and cardiovascular disease. Because single bouts of exercise are established to improve metabolic and vascular insulin sensitivity in people with obesity, the investigators anticipate exercise to raise brain insulin sensitivity in relation to cognition and cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >/=40 and </=80 years old.
* Has a body mass index >/=25 and </=45 kg/m2.
* Physical Activity (<150 min of moderate/high intensity exercise per week)

Exclusion Criteria:

* Subjects who have not been weight stable (>2 kg weight change in past 3 months)
* Subjects who are smokers or who have quit smoking <1 years ago
* Subjects with abnormal estimated glomerular filtration rate (eGFR).
* Hypertriglyceridemic (>400 mg/dl) and hypercholesterolemic (>260 mg/dl) subjects
* Hypertensive (>160/100 mmHg)
* Subjects with a history of significant metabolic, cardiac, congestive heart failure, cerebrovascular, hematological, pulmonary, gastrointestinal, liver, renal, or endocrine disease or cancer that in the investigator's opinion would interfere with or alter the outcome measures or impact subject safety.
* Pregnant (as evidenced by positive urine pregnancy test) or nursing women
* Subjects with contraindications to participation in an exercise
* Current Pregnancy
* Currently taking active weight suppression medication (e.g. phentermine, orlistat, lorcaserin, naltrexone-bupropion in combination, liraglutide, benzphetamine, diethylpropion, phendimetrazine)
* Subjects currently taking medications that affect heart rate and rhythm (i.e. Ca++ channel blockers, nitrates, alpha- or beta-blockers).
* Known contraindications for MRI imaging

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Brain insulin sensitivity | Change from baseline to exercise; about 1 week apart
  MRI arterial spin labeling, cerebral blood flow

SECONDARY OUTCOMES:
Cognition | Change from baseline to exercise; about 1 week apart
  NIH Toolbox Cognitive Battery
Blood Glucose | Change from baseline to exercise; about 1 week apart
  Blood draw via oxidase method
Blood Free Fatty Acids | Change from baseline to exercise; about 1 week apart
  Blood draw via colorimetric assays
Carbohydrate Use | Change from baseline to exercise; about 1 week apart
  Indirect Calorimetry
Systolic and Diastolic Blood Pressure | Change from baseline to exercise; about 1 week apart
  Cuff around arm

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Malin, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (4):
- United States (4):
  - Institute for Food, Nutrition, and Health, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Clinical Research Center, New Brunswick, New Jersey
  - Rutgers University Loree Gymnasium, New Brunswick, New Jersey
  - Center for Advanced Human Brain Imaging Research, Piscataway, New Jersey

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05853913/ICF_000.pdf